CLINICAL TRIAL: NCT04595318
Title: Feasibility and Preliminary Effectiveness of Varenicline for Co-occurring Cannabis and Tobacco Use
Brief Title: Varenicline for Co-occurring Cannabis and Tobacco Use
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2010-279-12; R25GM104547 (NIH); K23DA025736 (NIH); R25DA023021 (NIH)
Record Dates: First submitted 2016-04-28; First posted 2020-10-20 (Actual); Results first posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-08

CONDITIONS: Cannabis Dependence; Tobacco Dependence
MeSH Terms: conditions — Marijuana Abuse; Tobacco Use Disorder | interventions — Varenicline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | US Export: Yes

ARMS (2):
- Standard clinical care first, followed by standard clinical care and varenicline (Experimental): Four weeks of standard clinical care (SCC) in an outpatient substance use disorder treatment program. SCC includes individual counseling, at least once a month, that uses motivational and cognitive behavioral strategies, may address cannabis or tobacco use, and is delivered by trained substance use disorder treatment counselors; and medications for opioid use disorder (MOUD).
  This is followed by four weeks of SCC plus varenicline treatment (SCC and VT). Varenicline treatment included a gour-week supply of standard doses: 0.5mg for the first three days, 0.5mg twice a day for the following four days, and 1 mg twice a day for the remaining 21 days.
  Interventions: Drug: Standard clinical care first, followed by standard clinical care and varenicline
- Standard clinical care and varenicline first, followed by standard clinical care (Experimental): Four weeks of standard clinical care (SCC) plus varenicline treatment (SCC and VT). SCC includes individual counseling, at least once a month, that uses motivational and cognitive behavioral strategies, may address cannabis or tobacco use, and is delivered by trained substance use disorder treatment counselors; and medications for opioid use disorder (MOUD).Varenicline treatment included a gour-week supply of standard doses: 0.5mg for the first three days, 0.5mg twice a day for the following four days, and 1 mg twice a day for the remaining 21 days.
  This is followed by four weeks of SCC in an outpatient substance use disorder treatment program, as described above.
  Interventions: Drug: Standard clinical care and varenicline first, followed by standard clinical care

INTERVENTIONS:
Drug: Standard clinical care first, followed by standard clinical care and varenicline — Standard clinical care includes substance use disorder treatment program-based individual behavioral counseling at least once a month using motivational and cognitive behavioral strategies. Varenicline therapy includes a one month's supply of the medication in standard doses: 0.5 mg for 3 days, 0.5 mg twice a day for 4 days, then 1 mg twice a day for 21 days.
  Other Names: SCC first, then SCC+VT
  Arms: Standard clinical care first, followed by standard clinical care and varenicline
Drug: Standard clinical care and varenicline first, followed by standard clinical care — Standard clinical care includes substance use disorder treatment program-based individual behavioral counseling at least once a month using motivational and cognitive behavioral strategies. Varenicline therapy includes a one month's supply of the medication in standard doses: 0.5 mg for 3 days, 0.5 mg twice a day for 4 days, then 1 mg twice a day for 21 days.
  Other Names: SCC+VT first, then SCC
  Arms: Standard clinical care and varenicline first, followed by standard clinical care

SUMMARY:
Pilot, eight week, open-label, within-subject cross over trial of four weeks of standard clinical care (SCC) in an outpatient substance use disorder treatment program and four weeks of SCC and varenicline among current and former tobacco smokers with frequent cannabis use.

DETAILED DESCRIPTION:
Treating co-occurring cannabis and tobacco use disorders might reduce the health burdens associated with both substances. However, few studies have evaluated pharmacological interventions, in combination with behavioral treatment, to address co-occurring cannabis and tobacco use; these are limited by high participant attrition, poor adherence to interventions, and lack of control. Pilot, eight week, open-label, within-subject cross over trial of four weeks of standard clinical care (SCC) in an outpatient substance use disorder treatment program and four weeks of SCC and varenicline among current and former tobacco smokers with frequent cannabis use. Participants were recruited from an urban, outpatient substance use disorder treatment program that offers both intensive behavioral counseling and medications for opioid use disorder (MOUD). Participants were randomized to receive either SCC or SCC and varenicline first and then were crossed over to receive the opposite intervention. The study consisted of two 4-week treatment periods with no washout period. Outcomes are reported in pooled analyses of all participants in each treatment phase.

ELIGIBILITY:
Inclusion Criteria:

* Able to speak English
* Uses cannabis at least 5 days in the past 7 days
* Current or former tobacco smoker
* Has not taken varenicline in the past 30 days
* Not pregnant, trying to conceive or breastfeeding
* Able to provide informed consent
* Test positive for cannabinoids by urine toxicology

Exclusion Criteria:

* Unstable medical or psychiatric illness
* Opioid use disorder was initially exclusionary but eligibility criteria were revised after 32 individuals were screened to facilitate recruitment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shadi Nahvi, Principal Investigator — Montefiore Medical Center

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from an urban, outpatient substance abuse treatment program that offers both intensive behavioral counseling and medication-assisted treatment (MAT) for opioid use disorder. These clinical sites were selected based on being able to successfully recruit and retain participants during prior clinical trials along with an anticipation of high prevalence of persons with frequent cannabis use in the area.
Pre-assignment Details: 193 individuals in treatment at an outpatient substance use disorder treatment program were screened for eligibility. Of the 186 participants who were not enrolled and randomized, 182 were ineligible and 4 declined to participate. Seven participants were eligible and enrolled and randomized into the eight-week, open-label, within-subject cross over trial.
Groups:
- Standard Clinical Care (SCC) First, Followed by Standard Clinical Care and Varenicline (SCC and VT): Participants received four weeks of standard clinical care (SCC) in an outpatient substance use disorder treatment program. SCC included individual counseling, at least once a month, that used motivational and cognitive behavioral strategies, addressed cannabis or tobacco use, as needed, and was delivered by trained substance use disorder treatment counselors; and medications for opioid use disorder (MOUD).
  This was followed by four weeks of standard clinical care (SCC) plus varenicline treatment (SCC and VT). SCC included individual counseling, at least once a month, that used motivational and cognitive behavioral strategies, addressed cannabis or tobacco use, as needed, and was delivered by trained substance use disorder treatment counselors; and medications for opioid use disorder (MOUD).Varenicline treatment included a four-week supply of standard doses: 0.5mg for the first three days, 0.5mg twice a day for the following four days, and 1 mg twice a day for the remaining 21 days.
- Standard Clinical Care and Varenicline First (SCC + VT), Followed by Standard Clinical Care (SCC): Participants received four weeks of standard clinical care (SCC) plus varenicline treatment (SCC and VT). SCC included individual counseling, at least once a month, that used motivational and cognitive behavioral strategies, addressed cannabis or tobacco use, as needed, and was delivered by trained substance use disorder treatment counselors; and medications for opioid use disorder (MOUD).Varenicline treatment included a four-week supply of standard doses: 0.5mg for the first three days, 0.5mg twice a day for the following four days, and 1 mg twice a day for the remaining 21 days.
  This was followed by four weeks of standard clinical care (SCC) in an outpatient substance use disorder treatment program. SCC included individual counseling, at least once a month, that used motivational and cognitive behavioral strategies, addressed cannabis or tobacco use, as needed, and was delivered by trained substance use disorder treatment counselors; and medications for opioid use disorder (MOUD).
Period: First Intervention (Four Weeks)
Arm/Group | Standard Clinical Care (SCC) First, Followed by Standard Clinical Care and Varenicline (SCC and VT) | Standard Clinical Care and Varenicline First (SCC + VT), Followed by Standard Clinical Care (SCC)
Started | 3 (In a deviation from the trial design, one participant completed SCC alone for two weeks, then SCC+VT for four weeks, followed by SCC alone for two weeks.) | 4
Completed | 3 (In a deviation from the trial design, one participant completed SCC alone for two weeks, then SCC+VT for four weeks, followed by SCC alone for two weeks.) | 4
Not Completed | 0 | 0
Period: Second Intervention (Four Weeks)
Arm/Group | Standard Clinical Care (SCC) First, Followed by Standard Clinical Care and Varenicline (SCC and VT) | Standard Clinical Care and Varenicline First (SCC + VT), Followed by Standard Clinical Care (SCC)
Started | 3 | 4
Completed | 3 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: There were a total of 7 participants in the trial who were randomized to the sequence of intervention. All participants completed a sequence of 4 weeks of standard clinical care and standard clinical care plus varenicline in some order predicated on assignment in this crossover study design.
Groups:
- All Study Participants: Participants received either four weeks of standard clinical care (SCC) in an outpatient substance use disorder treatment program followed by four weeks of standard clinical care (SCC) plus varenicline treatment (SCC and VT) or four weeks of standard clinical care (SCC) plus varenicline treatment (SCC and VT) followed by four weeks of standard clinical care (SCC) in an outpatient substance use disorder treatment program as detailed in the Participant Flow Arm/Group Description
Arm/Group | All Study Participants
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Black or African American | 2
  Non-Hispanic White | 1
Region of Enrollment [Number; unit: participants]
  United States | 7
Cannabis Craving [Mean (Standard Deviation); unit: score on a scale] — Cannabis craving was assessed using the Marijuana Craving Questionnaire-Short Form (MCQ-SF) a self-reporting tool with 12 items rated on a 7-point Likert scale from 1 (strongly disagree) to 7 (strongly agree). The 12 items are grouped by certain characteristics and the score of each of resulting groups correlates to the intensity of the four craving dimensions (compulsivity, emotionality, expectancy, and purposefulness). Scores from the four subscales are summed with total possible scores ranging from 12 - 84. Higher scores are indicative of increased craving.
  score on a scale | 43 (20)
Cannabis Withdrawal [Mean (Standard Deviation); unit: score on a scale] — Cannabis withdrawal was measured by the 15-item version of the Marijuana Withdrawal Checklist (MWC). Participants rated each symptom experienced during their most recent period of marijuana abstinence, based on a 4-point scale where 0 = none, 1 = mild, 2 = moderate, and 3 = severe. A total MWC score was obtained by summing the responses. Possible total scoring ranges from 0 - 45, with 0 signifying no withdrawal symptoms and 45 signifying the most severe withdrawal symptoms.
  score on a scale | 10 (11)
Quantity of Cannabis Use [Number; unit: percentage of days] — The quantity of cannabis use was measured using the Timeline Follow-Back (TLFB) method. TLFB is a method in which participants use a physical calendar to quantify the number of days over a specified period of time (in this study 14 days) during which cannabis was used. An aggregate value for percentage of days of cannabis use was calculated for all study participants by tabulating the total number of days cannabis was actually used by all study participants over the prior 14-day period and dividing by the total number of calendar days over the period for the 7 participants (i.e., 14x7=98).
  percentage of days | 77
Frequency of Cannabis Use [Mean (Standard Deviation); unit: Cannabis use per day] — The frequency of cannabis use per day was evaluated over the prior 14-day period using the Timeline Follow-Back method (TLFB), a method in which participants used a physical calendar to self-report the number times per days cannabis was used.
  Cannabis use per day | 4 (0.5)
Number of Cigarettes Smoked Per Day [Mean (Standard Deviation); unit: Cigarettes smoked per day] — The number of cigarettes smoked per day was measured using Timeline Follow-Back (TLFB). TLFB is a method in which participants used a physical calendar to self-report the number of cigarettes smoked per day over the prior 14-day period in order to evaluate ongoing tobacco usage.
  Cigarettes smoked per day | 13 (9)
Number of participants with Toxicology-verified cannabis abstinence [Count of Participants; unit: Participants] — The number of participants with Toxicology-verified cannabis abstinence was determined by applying the TLFB method and then biochemically confirming the number of participants with a urine tetrahydrocannabinol (THC) levels less than 50 ng/ml.
  Participants | 1
Number of participants with biochemically-verified tobacco abstinence [Count of Participants; unit: Participants] — The number of participants with biochemically-verified tobacco abstinence was determined by applying the TLFB method and then biochemically verified by measuring participant levels of expired carbon monoxide < 8 parts per million (CO < 8ppm). The Bedfont Smokerlyzer carbon monoxide monitor was used in the analysis.
  Participants | 1
Mean expired carbon monoxide (CO) [Mean (Standard Deviation); unit: parts per million (ppm)] — Mean expired carbon monoxide (CO) per participant was measured using the Bedfont Smokerlyzer carbon monoxide monitor. Results reported in mean parts per million (ppm)
  parts per million (ppm) | 9 (6)

OUTCOME MEASURES:

1. Primary Outcome: Enrollment Rate
Description: Percentage of the eleven eligible subjects willing to participate
Time Frame: Baseline
Population: In a deviation from the trial design, one participant completed SCC alone for two weeks, then SCC+VT for four weeks, followed by SCC alone for two weeks.
Measure: Count of Participants; unit: Participants
Groups:
- All Study Participants: Participants received four weeks of standard clinical care (SCC) in an outpatient substance use disorder treatment program. SCC included individual counseling, at least once a month, that used motivational and cognitive behavioral strategies, addressed cannabis or tobacco use, as needed, and was delivered by trained substance use disorder treatment counselors; and medications for opioid use disorder (MOUD).
  Participants also received four weeks of SCC plus varenicline treatment (SCC+VT). Varenicline treatment included a four-week supply of standard doses: 0.5mg for the first three days, 0.5mg twice a day for the following four days, and 1 mg twice a day for the remaining 21 days.
  Of the 7 participants on study, three participants were randomized to begin with four weeks of SCC followed by four weeks of SCC+VT and four participants were randomized to begin with four weeks of SCC+VT followed by four weeks of SCC only.
Arm/Group | All Study Participants
Number analyzed (Participants) | 11
Participants | 7

2. Secondary Outcome: Retention Rate
Description: Retention rate was determined by the percentage of participants who completed all study visits.
Time Frame: Week 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 7
Participants | 7

3. Secondary Outcome: Overall Medication Adherence
Description: Overall medication adherence was calculated as a percentage based on the number of pills prescribed during the study, corrected for the number of pills returned, divided by the period (in days), and multiplied by 100. An aggregate percentage of pills was calculated and reported for all seven study participants.
Time Frame: Upon conclusion of SCC+Varenicline treatment (4 weeks or 8 weeks based on randomization to arm/group)
Population: as for outcome 1
Measure: Number; unit: Percentage of pills
Arm/Group | All Study Participants
Number analyzed (Participants) | 7
Percentage of pills | 62

4. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events: Upset Stomach
Description: The number of participants with a self-reported adverse event of upset stomach was determined using a structured questionnaire of common varenicline symptoms
Time Frame: Upon conclusion of SCC+VT treatment (4 weeks or 8 weeks based on randomization to arm/group)
Population: While receiving standard clinical care without Varenicline participants were not assessed for Varenicline associated adverse effects. In a deviation from the trial design, one participant completed SCC alone for two weeks, then SCC+VT for four weeks, followed by SCC alone for two weeks.
Measure: Number; unit: participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 7
participants | 5

5. Secondary Outcome: Number of Participants With Treatment-Emergent Symptoms of Major Depressive Disorder
Description: The number of participants with self-reported Treatment-Emergent symptoms of major depressive disorder was determined using the MINI International Neuropsychiatric Interview (M.I.N.I), a short structured diagnostic interview tool used to assess DSM-IV and ICD-10 psychiatric disorders
Time Frame: Upon conclusion of SCC+VT treatment (4 weeks or 8 weeks based on randomization to arm/group)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 7
Participants | 1

6. Secondary Outcome: Cannabis Craving
Description: Cannabis craving was assessed using the Marijuana Craving Questionnaire-Short Form (MCQ-SF). The MCQ-SF is a valid and reliable, self-report instrument with 12 items rated on a 7-point Likert scale from 1 (strongly disagree) to 7 (strongly agree). The 12 items are grouped by certain characteristics and the score of each of resulting groups correlates to the intensity of the four craving dimensions (compulsivity, emotionality, expectancy, and purposefulness). Scores from the four subscales are summed with total possible scores ranging from 12 - 84. Higher scores are indicative of increased craving.
Time Frame: Week 4 and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Study Participants
Number analyzed (Participants) | 7
score on a scale
  SCC | 34 (20)
  SCC+VT | 35 (23)

7. Secondary Outcome: Cannabis Withdrawal
Description: Cannabis withdrawal was measured by the 15-item version of the Marijuana Withdrawal Checklist (MWC). Participants rated each symptom experienced during their most recent period of marijuana abstinence, based on a 4-point scale where 0 = none, 1 = mild, 2 = moderate, and 3 = severe. A total MWC score was obtained by summing the responses. Possible total scoring ranges from 0 - 45, with 0 signifying no withdrawal symptoms and 45 signifying the most severe withdrawal symptoms.
Time Frame: Week 4 and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Study Participants
Number analyzed (Participants) | 7
score on a scale
  SCC | 4 (6)
  SCC+VT | 4 (5)

8. Secondary Outcome: Quantity of Cannabis Use
Description: The quantity of cannabis use over the prior 14-day period was measured using the Timeline Follow-Back (TLFB) method. TLFS is a method in which participants used a physical calendar to quantify the number of days over a specified period of time (in this study 14 days) during which cannabis was used. An aggregate value for percentage of days of cannabis use was calculated by tabulating the total number of days cannabis was used by all study participants over the prior 14-day period and dividing by the total number of calendar days over this period across the 7 participants (i.e., 14x7=98).
Time Frame: Week 4 and Week 8
Population: as for outcome 1
Measure: Number; unit: percentage of days
Arm/Group | All Study Participants
Number analyzed (Participants) | 7
percentage of days
  SCC | 82
  SCC+VT | 60

9. Secondary Outcome: Frequency of Cannabis Use
Description: The frequency of cannabis use per day was evaluated over the prior 14-day period using the Timeline Follow-Back method (TLFB), a method in which participants used a physical calendar to self-report the number times per days cannabis was used.
Time Frame: Week 4 and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Cannabis use per day
Arm/Group | All Study Participants
Number analyzed (Participants) | 7
Cannabis use per day
  SCC | 3 (0.4)
  SCC+VT | 2 (0.3)

10. Secondary Outcome: Number of Cigarettes Smoked Per Day
Description: The number of cigarettes smoked per day was measured using Timeline Follow-Back (TLFB). TLFB is a method in which participants used a physical calendar to self-report the number of cigarettes smoked per day over the prior 14-day period in order to evaluate ongoing tobacco usage.
Time Frame: Week 4 and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Cigarettes smoked per day
Arm/Group | All Study Participants
Number analyzed (Participants) | 7
Cigarettes smoked per day
  SCC | 5 (7)
  SCC+VT | 5 (7)

11. Secondary Outcome: Number of Participants With Toxicology-verified Cannabis Abstinence
Description: The number of participants with Toxicology-verified cannabis abstinence was determined by applying the TLFB method and then biochemically confirming the number of participants with a urine tetrahydrocannabinol (THC) levels less than 50 ng/ml.
Time Frame: Week 4 and Week 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 7
Participants
  SCC | 1
  SCC+VT | 1

12. Secondary Outcome: Number of Participants With Biochemically-verified Tobacco Abstinence
Description: The number of participants with biochemically-verified tobacco abstinence was determined by applying the TLFB method and then biochemically verified by measuring participant levels of expired carbon monoxide < 8 parts per million (CO < 8ppm). The Bedfont Smokerlyzer carbon monoxide monitor was used in the analysis.
Time Frame: Week 4 and Week 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 7
Participants
  SCC | 2
  SCC+VT | 1

13. Secondary Outcome: Mean Expired Carbon Monoxide
Description: Mean expired carbon monoxide (CO) per participant was measured using the Bedfont Smokerlyzer carbon monoxide monitor. Results reported in mean parts per million (ppm)
Time Frame: Week 4 and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: parts per million (ppm)
Arm/Group | All Study Participants
Number analyzed (Participants) | 7
parts per million (ppm)
  SCC | 13 (9)
  SCC+VT | 14 (11)

14. Secondary Outcome: Number of Participants With Treatment-Emergent Suicidal Ideation Events
Description: The number of participants with treatment-emergent suicidal ideation events was determined using the Columbia Suicide Severity Rating Scale (C-SSRS). The C-SSRS contains 6 "yes" or "no" questions in which respondents are asked to indicate whether they have experienced several thoughts or feelings relating to suicide over the past month and behaviors over their lifetime as well as during the past 3 months. An answer of "yes" to any of the six questions may indicate a need for referral to a trained mental health professional and an answer of "yes" to questions to the final three questions indicates high-risk.
Time Frame: Week 4 and Week 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 7
Participants
  SCC | 0
  SCC+VT | 0

ADVERSE EVENTS:
Time Frame: Week 4 and Week 8
Groups:
- Standard Clinical Care (SCC ): Participants received four weeks of standard clinical care (SCC) in an outpatient substance use disorder treatment program. SCC included individual counseling, at least once a month, that used motivational and cognitive behavioral strategies, addressed cannabis or tobacco use, as needed, and was delivered by trained substance use disorder treatment counselors; and medications for opioid use disorder (MOUD).
- Standard Clinical Care and Varenicline (SCC + VT): Participants received four weeks of standard clinical care (SCC) plus varenicline treatment (SCC and VT). SCC included individual counseling, at least once a month, that used motivational and cognitive behavioral strategies, addressed cannabis or tobacco use, as needed, and was delivered by trained substance use disorder treatment counselors; and medications for opioid use disorder (MOUD).Varenicline treatment included a four-week supply of standard doses: 0.5mg for the first three days, 0.5mg twice a day for the following four days, and 1 mg twice a day for the remaining 21 days.
Arm/Group | Standard Clinical Care (SCC ) | Standard Clinical Care and Varenicline (SCC + VT)
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 5/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Clinical Care (SCC ) (N=7) | Standard Clinical Care and Varenicline (SCC + VT) (N=7)
insomnia (Nervous system disorders) | 0 (0) | 4 (4)
upset stomach (Gastrointestinal disorders) | 0 (0) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No